CLINICAL TRIAL: NCT04097587
Title: Parental Educational Intervention Reduces Screen Time and Improves Sleep Disturbances and Attention Problems in Preschool Children: a Clustered Randomized Controlled Study
Brief Title: Parental Education and Children's Screen Time
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Su-Ru Chen, Associate professor, Taipei Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: (TMU-JIRB N201803013)
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-09

CONDITIONS: Screen Time
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A clustered randomized controlled study with a parallel-group design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- control group (Other): received standard school classes and usual activities offered at the kindergarten. Briefly, kindergarten activities included daily learning activities, outdoor activities, breakfast, lunch, snacks, and nap time.
  Interventions: Behavioral: experimental group; Other: control group

INTERVENTIONS:
Behavioral: experimental group — This program was carried out for 50 min/week over 8 weeks to empower parents with knowledge and self-efficacy about children's screen use, and motivate them to monitor and change their children's screen behaviors. Teaching strategies included lectures, group discussions, reflection, role playing, and peer sharing (Table 1). Topics included 1) parents' and children's screen use, 2) the relationship between network equipment and children's internet use, 3) the positive and negative effects of excessive screen use on children's physical and psychological development, 4) limiting screen use at mealtimes and bedtime, 5) strategies for screen-related devices, 6) alternative activities to screen use, such as board games and outdoor activities, 7) setting a target of appropriate screen times, and 8) encouraging the signing of a contract between parents and children to limit screen time. We also provided parents with a handbook of the course content.
  Other Names: parental educational program
Other: control group — received standard school classes and usual activities offered at the kindergarten. Briefly, kindergarten activities included daily learning activities, outdoor activities, breakfast, lunch, snacks, and nap time.
  Other Names: usual activity

SUMMARY:
The study was to investigate the efficacy of a parental educational program on reducing screen use, and improving sleep quality and psychosocial adaptations in children aged 4-6 years.

DETAILED DESCRIPTION:
A total of 129 parent-child dyads were randomly allocated to two groups: experimental group (receiving parental education, n=63), and control group (daily activities, n=66). Data were collected before and after intervention. Instruments included screen time, Children's Sleep Habits Questionnaire, and Pediatric Symptom Checklist-17. A linear mixed model analysis was used to examine the efficacy of education intervention.

ELIGIBILITY:
Inclusion Criteria:

* children aged 4~6 years with screen time of ≥ 2 h/day.

Exclusion Criteria:

* cerebral palsy,
* mental retardation
* psychosis
* Down's syndrome
* chronic disease
* hearing impairment.

Ages: 48 Months to 72 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2018-12-28 (Actual)

PRIMARY OUTCOMES:
screen time | one week assessment
  children's screen time, was measured by parents as the time children spent watching TV/DVD/videos, playing TV games, and using a computer on weekdays and weekends.

CONTACTS AND LOCATIONS:
Locations (1):
- Su-Ru Chen, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zhao J, Zhang Y, Jiang F, Ip P, Ho FKW, Zhang Y, Huang H. Excessive Screen Time and Psychosocial Well-Being: The Mediating Role of Body Mass Index, Sleep Duration, and Parent-Child Interaction. J Pediatr. 2018 Nov;202:157-162.e1. doi: 10.1016/j.jpeds.2018.06.029. Epub 2018 Aug 9. PMID 30100232
- See also: reference link — https://www.ncbi.nlm.nih.gov/pubmed/30100232